CLINICAL TRIAL: NCT03688425
Title: Clinical Study to Compare Clinical Outcomes of Trifocal IOLs FineVision POD L GF and FineVision POD F GF After Bilateral Implantation in Asian Eyes
Brief Title: Comparison of Clinical Outcomes POD L GF vs POD F GF in Asian Eyes
Acronym: PHY1802
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHY1802
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Cataract; Lens Opacities; Presbyopia
Keywords: Intraocular Lens; trifocal; hydrophobic
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOL implantation experimental (Experimental): hydrophobic, trifocal intraocular lens POD L GF with light distribution far > intermediate > near
  Interventions: Device: IOL implantation experimental
- IOL implantation active comparator (Active Comparator): hydrophobic, trifocal intraocular lens POD F GF with light distribution far > near > intermediate
  Interventions: Device: IOL implantation active comparator

INTERVENTIONS:
Device: IOL implantation experimental — Implantation of trifocal IOL POD F GF consisting of light distribution order: far > intermediate > near
  Arms: IOL implantation experimental
Device: IOL implantation active comparator — Implantation of trifocal IOL POD F GF consisting of light distribution order: far > near > intermediate
  Arms: IOL implantation active comparator

SUMMARY:
Prospective, randomised, controlled, single-surgeon, single-center clinical study to compare the clinical outcomes of two trifocal IOLs differing in the dominance of additional power. The investigational device POD L GF shows dominance for the intermediate addition (+1.75 D), whereas the control device POD F GF shows dominance for the near addition (+3.5 D). Implantation of the IOLs is bilaterally.

DETAILED DESCRIPTION:
This is a prospective, randomised, controlled, single-surgeon, single-center clinical study whereby patients undergoing routine cataract surgery will have bilateral implantation of trifocal intraocular lenses. The patients will either be implanted with the hydrophobic IOL FineVision POD L GF or the hydrophobic IOL FineVision POD F GF (both lenses: (PhysIOL, Liège, Belgium).

The devices under investigation (FineVision POD L GF and POD F GF) are trifocal glistening-free acrylic intraocular lenses (IOLs) manufactured by the sponsor of this study PhysIOL sa/nv. Both consist of the same hydrophobic material. The main difference between the lenses is the dominance of additional power. The investigational device POD L GF shows dominance for the intermediate addition (+1.75 D), whereas the control device POD F GF shows dominance for the near addition (+3.5 D). The IOLs will be implanted as part of the routine cataract surgery on patients suffering from cataract development.

Subjects participating in the trial will attend a total of 10 study visits (1 preoperative, 2 operative and 7 postoperative) over a period of 6 months. Subjects would have the option for unscheduled visits if required medically.

Primary and secondary endpoint data will be collected at the 6 months follow up visit. Data analyses will be done after the last patient finished the final examination to support the study publication plan.

ELIGIBILITY:
Inclusion Criteria:

* Cataractous eyes with no comorbidity
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent

Exclusion Criteria:

* Age of patient <40 years
* Irregular astigmatism
* Regular corneal astigmatism >0.75 dioptres by an automatic keratometer or biometer or >1.0 dioptres if the steep axis of cylinder is between 90° and 120°
* Difficulty for cooperation (distance from their home, general health condition)
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus (with retinopathy), immunocompromised, glaucoma etc…)
* Any ocular comorbidity
* History of ocular trauma or prior ocular surgery including refractive procedures
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, chronic Uveitis, Marfan's syndrome)
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions)
* AMD suspicious eyes (determined by OCT)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
monocular Best Corrected Distance Visual Acuity (CDVA) under photopic light conditions. | 3 months postoperative
  No statistically significant difference between the two study groups on monocular CDVA at 3 months follow up visit. A significance level of 0.05 or lower (p < 0.05) will be considered statistically significant. CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2014.

SECONDARY OUTCOMES:
Manifested refraction | 3 months postoperative
  The manifested refraction is measured by means of a phoropter. The data contains values for sphere, cylinder and axis of cylinder according to ISO 11979-7:2014. This data will also be used to calculate the manifested refractive spherical equivalent (MRSE)
Uncorrected Distance Visual Acuity (UDVA) under photopic light conditions | 3 months postoperative
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014. This assessment is done monocularly and binocularly under photopic light conditions.
Uncorrected Distance Visual Acuity (UDVA) under mesopic light conditions | 6 months postoperative
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014. This assessment is done monocularly under mesopic light conditions.
Corrected Distance Visual Acuity (CDVA) under photopic light conditions | 3 months postoperative
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2014. This assessment is done binocularly under photopic light conditions.
Corrected Distance Visual Acuity (CDVA) under mesopic light conditions | 6 months postoperative
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2014. This assessment is done monocularly under mesopic light conditions.
Distance Corrected Intermediate Visual Acuity at 70cm (DCIVA) under photopic light conditions | 3 months postoperative
  DCIVA is measured with ETDRS charts placed in 70cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly and binocularly under photopic light conditions.
Distance Corrected Intermediate Visual Acuity at 70cm (DCIVA) under mesopic light conditions | 6 months postoperative
  DCIVA is measured with ETDRS charts placed in 70cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly under mesopic light conditions.
Uncorrected Intermediate Visual Acuity at 70cm (UIVA) under photopic light conditions | 3 months postoperative
  UIVA is measured with ETDRS charts placed in 70cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done monocularly and binocularly under photopic light conditions.
Uncorrected Intermediate Visual Acuity at 70cm (UIVA) under mesopic light conditions | 6 months postoperative
  UIVA is measured with ETDRS charts placed in 70cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done monocularly under mesopic light conditions.
Distance Corrected Near Visual Acuity at 35cm (DCNVA) under photopic light conditions | 3 months postoperative
  DCNVA is measured with ETDRS charts placed in 35cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly and binocularly under photopic light conditions.
Distance Corrected Near Visual Acuity at 35cm (DCNVA) under mesopic light conditions | 6 months postoperative
  DCNVA is measured with ETDRS charts placed in 35cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly under mesopic light conditions.
Uncorrected Near Visual Acuity at 35cm (UNVA) under photopic light conditions | 3 months postoperative
  UNVA is measured with ETDRS charts placed in 35cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done monocularly and binocularly under photopic light conditions.
Uncorrected Near Visual Acuity at 35cm (UNVA) under mesopic light conditions | 6 months postoperative
  UNVA is measured with ETDRS charts placed in 35cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done monocularly under mesopic light conditions.
Contrast Sensitivity | 3 months postoperative
  Contrast Sensitivity under photopic and mesopic light conditions
Aberrometry | 3 months postoperative
  Aberrometry outcomes are measured with a standard aberrometer. The following values will be evaluated in this study: Spherical aberrations, high order aberrations, lens tilt.
AcuTarget diagnostic device | 3 months postoperative
  Measurement of Ocular Scatter Index (OSI) score to evaluate and compare the scattering of the implanted lenses.
Questionnaire VFQ-25 (National Eye Institute) | 3 months postoperative
  Outcomes measures of a questionnaire to address the general patient satisfaction and possible side effects of the treatment. For this study, the validated and verified questionnaire VFQ-25 (National Eye Institute) will be used. The maximum score for each question is 100.
Defocus Curve monocular | 1 month postoperative
  To assess the visual acuity for different distances, defocus curves under photopic light conditions are measured. This test is performed with best distance corrected refraction and spherical additions ranging from -5.0 D to +1.5 D. This examination is performed monocularly.
Defocus Curve binocular | 3 months postoperative
  To assess the visual acuity for different distances, defocus curves under photopic light conditions are measured. This test is performed with best distance corrected refraction and spherical additions ranging from -5.0 D to +1.5 D. This examination is performed binocularly.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Edward Ang, MD, Principal Investigator — Asian Eye Institute
Locations (1):
- Asian Eye Institute, Makati City, Philippines

IPD SHARING:
Plan to Share IPD: No